CLINICAL TRIAL: NCT04915222
Title: Comparison Between the Effectiveness of Manual Cervical Traction and Natural Apophyseal Glides on Pain and Disability Among Patients With Cervical Radiculopathy
Brief Title: Manual Cervical Traction and Natural Apophyseal Glides for Cervical Radiculopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Mariam Ghazanfar, Senior Lecturer, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 129/RC/KEMU
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical radiculopathy; manual traction; neck pain
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Intervention Model Description: Single center, parallel group randomized controlled trial of 72 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural apophyseal glides (Experimental): This group receives natural apophyseal glides along with conventional physical therapy and manual techniques as treatment for 3 sessions per week on alternate days for 3 weeks
  Interventions: Other: Natural apophyseal glides
- Cervical manual traction (Active Comparator): This group receives cervical manual traction along with conventional physical therapy and manual techniques as treatment for 3 sessions per week on alternate days for 3 weeks
  Interventions: Other: Cervical manual traction

INTERVENTIONS:
Other: Natural apophyseal glides — Patients received conventional therapy and NAGS with 2-3 hertz (less than 6 repetitions) in 3 sets for 3 weeks. The conventional therapy included hot pack, Neck range of motion exercises, neck strengthening and stabilization exercises. The hot pack is a form of thermo therapywas applied for 10 to 15 minutes and was applied at each visit during 3 sessions per week for total 3 weeks. The strengthening and stabilization exercises are form of therapeutics exercise are prescribed at 15 to 20 times per session for total 3 weeks. Intensity of exercise may rise gradually according to patient tolerance and muscular strength.
  Arms: Natural apophyseal glides
Other: Cervical manual traction — Patients received cervical manual traction (CMT) along with traditional therapy. Treatment frequency was 3 sessions per week for total three weeks duration. CMT applied was intermittent type traction.8 to 10 kg force was applied at an angle of 20 to 25 degree from horizontal. 5sets of cervical traction are performed. In every set traction is given for 1 minute with rest period of 20 seconds. The total time of traction session was 10 minute. The conventional therapy included hot pack, Neck range of motion exercises, neck strengthening and stabilization exercises. The hot pack is a form of thermo therapywas applied for 10 to 15 minutes and was applied at each visit during 3 sessions per week for total 3 weeks. The strengthening and stabilization exercises are form of therapeutics exercise are prescribed at 15 to 20 times per session for total 3 weeks. Intensity of exercise may rise gradually according to patient tolerance and muscular strength.
  Arms: Cervical manual traction

SUMMARY:
Cervical Radiculopathy is a clinical disorder of nerve root, and often is due to compressive or inflammatory pathology. There are number of different procedures which have been suggested for decreasing pain and disability in patients but manual therapy has been validated the effective technique. The objective of current research was to assess the comparative effectiveness of the Manual Cervical Traction and the Natural Apophyseal Glides on pain and disability among Cervical Radiculopathy patients.

A parallel design, randomized controlled trial was performed on 72 patients in physiotherapy department, Mayo Hospital Lahore. Participants were randomly allocated into two groups after baseline testing. Group A received natural apophyseal glides and baseline treatment and group B received manual cervical traction and baseline treatment. Treatment period was of 3 weeks with 3 weekly sessions on alternate basis. Assessment was done before treatment at baseline and then by second and third week using numeric pain rating scale and neck disability index. SPSS version 25 was used to analyzed the data.

DETAILED DESCRIPTION:
72 patients who fulfill the inclusion criteria were enrolled in this study. Written informed consent was taken from every subject participating in this study. Allocation of subjects in two groups has been done by random number table as per CONSORT guidelines 2010. Group A was treated with Natural Apophyseal Glides and group B with Manual Cervical Traction. Both groups received the conventional therapy along with the manual techniques. The conventional therapy included hot pack, Neck range of motion exercises, neck strengthening and stabilization exercises. The hot pack is a form of thermo therapywas applied for 10 to 15 minutes and was applied at each visit during 3 sessions per week for total 3 weeks. The strengthening and stabilization exercises are form of therapeutics exercise are prescribed at 15 to 20 times per session for total 3 weeks. Intensity of exercise may rise gradually according to patient tolerance and muscular strength.The conventional or baseline therapy remained same throughout the study.

Group A received conventional therapy and NAGS with 2-3 hertz (less than 6 repetitions) in 3 sets for 3 weeks. Group B received MCT along with traditional therapy. Treatment frequency was 3 sessions per week for total three weeks duration. MCT applied was intermittent type traction.8 to 10 kg force was applied at an angle of 20 to 25 degree from horizontal. 5sets of cervical traction are performed. In every set traction is given for 1 minute with rest period of 20 seconds. The total time of session was 10 minute.Pain intensity was measured by Numeric Pain Rating Scale. Functional ability was appraised by Neck Disability Index. All the information was collected by using standardized questionnaire of NPRS and NDI. Confounding variables are controlled by randomization and restriction methods. All treatment was given by single handed to control the biasness.Proforma of the patients which dropout during study was filled through intention to treat analysis method which was set as 15%.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically and radiologically diagnosed cervical radicular disease
* Subjects with difficulties in carrying out daily activities due to radicular pain
* Subject with bilateral/unilateral or both radicular pain
* Both male, female patients between 20 and 60 years with the radicular pain

Exclusion Criteria:

* Subjects having the mechanical cervical pain or the nonspecific pain of neck
* Subjects having cervical myelopathy
* Patients having any spine surgery or any malignancy
* Subjects having pain because of postural imbalances

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Numeric Pain Rating Scale | Baseline and 3 weeks
  Pain intensity was measured using numeric pain rating scale
Change from Baseline in Neck Disability Index | Baseline and 3 weeks
  Functional ability was measured using neck disability index

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Ghazanfar, Principal Investigator — University of Lahore
Locations (1):
- Physiotherapy Department of Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data